CLINICAL TRIAL: NCT04442009
Title: Ultrasound-guided Superficial Cervical Plexus Block for Pain Management After Orthognathic Surgery.
Brief Title: Superficial Cervical Plexus Block for Orthognathic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 15
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Maxillofacial Injuries; Maxillofacial Trauma; Maxillofacial Abnormalities; Maxillofacial Dysostosis
Keywords: Orthognathic surgery; Postoperative pain management; Superficial cervical plexus block
MeSH Terms: conditions — Maxillofacial Injuries; Maxillofacial Abnormalities; Maxillofacial Dysostosis

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is superficial cervical plexus block group. The second one is no intervention control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S = SCPB group (Active Comparator): US-guided SCPB will be performed at the end of the surgery before extubation, with patients in the supine position by using US (Vivid Q, GE Healthcare, US). Under aseptic conditions using 10% povidone iodine, the high frequency linear probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath and a 22G, 50 mm block needle (Braun Stimuplex Ultra 360, Germany) will be used.
  Sternocleidomastoid (SCM) muscle will be visualized. The 22 G needle will be inserted between the SCM and the prevertebral fascia by using in plane technique horizontally. The needle tip will be corrected with injecting 2 ml of normal saline. Then a 20 mL dose of 0.25% bupivacaine will be injected here. The same procedure will be performed for the opposite site (totally 40 mL dose of 0.25% bupivacaine).
  Interventions: Other: Group SCPB
- Group C = Control group (No Intervention): Patients will be administered dexketoprofen 50 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.

INTERVENTIONS:
Other: Group SCPB — In group SCBP, SCBP block will be performed. Patients will be administered dexketoprofen 50 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.
  Arms: Group S = SCPB group

SUMMARY:
US-guided superficial cervical plexus block (SCPB) may be used for several head and neck surgeries. Local anesthetic is injected under the sternocleidomastoid muscle for SCPB. It has lower complication rate compared to the deep cervical plexus block. Postoperative pain management is important in patients underwent orthognathic surgery. Effective pain treatment provides early mobilization, and shorter hospital stay.

DETAILED DESCRIPTION:
Postoperative pain management is very important in patients underwent orthognathic surgery. Effective pain control provides early mobilization, shorter hospital stay and it increases the satisfaction of the patients. Opioid agents may provide effective pain management, however opioid agents have undesirable adverse effects such as respiratory depression, sedation, constipation, nausea and vomiting etc. Ultrasound (US) -guided regional anesthesia techniques may be preferred for pain management in patients underwent orthognathic surgery. Regional anesthesia techniques may provide effective postoperative pain management as a part of multimodal analgesia regimens. US-guided bilateral superficial cervical plexus block (SCPB) have been performed for several head and neck surgeries and it provides effective pain control. The cervical plexus presents between the longus capitis and middle scalene muscles, under the prevertebral fascia. It is formed by the C2-4 cervical spinal nerves. There are the end points of these nerves in the interfascial area under the SCM. Thus, the superfascial branches of the cervical plexus may be blocked by injecting local anesthetic under the SCM. Cervical plexus may be blocked with deep or superficial technique. The deep CPB is defined as a paravertebral block. The deep branches may be targeted by this method. However it has some major disadvantages such as intravascular injection, epidural or subarachnoid injection, and phrenic nerve palsy, due to the deepness of the injection. Otherwise; SCPB is a superficial method and it has lower complication rate compared to the deep CPB. In an anatomical study, it has been reported that with SCPB there was spread of dye into the deep cervical fascia. The authors emphasized that this mechanism may explain the efficacy of the SCPB. Thus, with the SCPB both the superficial branches and the deep nerve roots may be blocked. Therefore, SCPB may provide effective pain management following orthognathic surgery. In the literature, there are no randomized clinical studies about pain management with US-guided SCPB after orthognathic surgery, yet.

The aim of this study is to evaluate the efficacy of the US-guided SCPB for postoperative analgesia management after orthognathic surgery. The primary aim is to evaluate postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting) compared to no intervention control group.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for orthognathic surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Change from baseline opioid consumption at postoperative 1, 2, 4, 8, 16, and 24 hours
  The primary aim is to compare postoperative opioid consumption

SECONDARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16, and 24 hours.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Kim JS, Ko JS, Bang S, Kim H, Lee SY. Cervical plexus block. Korean J Anesthesiol. 2018 Aug;71(4):274-288. doi: 10.4097/kja.d.18.00143. Epub 2018 Jul 4. PMID 29969890
- [Background] Raschke GF, Meissner W, Peisker A, Djedovic G, Rieger U, Guentsch A, Dammeier MG, Schultze-Mosgau S. Bilateral sagittal split osteotomy-parameters and correlations of postoperative pain management. Clin Oral Investig. 2018 Jan;22(1):181-187. doi: 10.1007/s00784-017-2097-z. Epub 2017 Mar 14. PMID 28293792
- [Background] Pandit JJ, Dutta D, Morris JF. Spread of injectate with superficial cervical plexus block in humans: an anatomical study. Br J Anaesth. 2003 Nov;91(5):733-5. doi: 10.1093/bja/aeg250. PMID 14570798